CLINICAL TRIAL: NCT03589599
Title: Understanding Tobacco Flavor Effects on Waterpipe Smokers' Experiences and Exposures
Brief Title: Understanding the Effect of Flavor on Hookah Smoking Experience
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida International University (Other)
Responsible Party: Principal Investigator, Wasim Maziak, phd, Professor and Chair, Department of Epidemiology, Florida International University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: R01DA042477 (NIH)
Record Dates: First submitted 2018-06-11; First posted 2018-07-18 (Actual); Last update posted 2020-08-03 (Actual); Status verified 2020-07

CONDITIONS: Waterpipe Smoking
MeSH Terms: conditions — Water Pipe Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Flavored tobacco (Experimental): All participants will be completing a lab visit where they smoke flavored waterpipe tobacco ad lib for up to 45 min.
  Interventions: Other: Flavored tobacco
- Non-flavored tobacco (Experimental): All participants will be completing a lab visit where they smoke non-flavored waterpipe tobacco ad lib for up to 45 min.
  Interventions: Other: Non-flavored tobacco

INTERVENTIONS:
Other: Flavored tobacco — Effects of flavored tobacco
  Arms: Flavored tobacco
Other: Non-flavored tobacco — Effects of non-flavored tobacco
  Arms: Non-flavored tobacco

SUMMARY:
This project addresses the need for evidence about the effect of flavoring manipulation on waterpipe smokers' satisfaction, dependence, harm perception, and toxicants exposure. Specifically, in this clinical study investigators will compare the effect on flavored and non-flavored waterpipe tobacco on smoking behavior, subjective experiences and toxicant exposure among waterpipe users. Findings from this study will help informing flavor-based product regulation by the FDA.

DETAILED DESCRIPTION:
Waterpipe (WP) tobacco smoking (a.k.a. hookah, shisha, narghile) is increasing rapidly in the United States (US), particularly among young people. Evidence suggests that WP smoking can lead to dependence, other tobacco use, and many of the known smoking-related diseases including cancer, cardiovascular disease and adverse pregnancy outcomes. These alarming trends led the Food and Drug Administration (FDA) in 2014 to propose including the WP under its regulatory authority, allowing the FDA to apply evidence-based regulatory approaches to control WP spread in the US. Given the salience of flavored tobacco in shaping the "WP experience", regulating WP tobacco flavor represents a promising approach for the FDA to curb WP use among US youth. This project aims to assist the FDA in these efforts by providing answers to specific questions pertinent to the potential of WP regulation through flavor. These include: - How would flavor manipulation affect the smoking experience and satisfaction of WP users at different stages of their smoking trajectory - How would smoking non-preferred flavor or unflavored WP tobacco reflects on smokers' exposure to nicotine, and dependence; and - How would flavor manipulation influence puffing behavior and exposure to toxicants such as carbon monoxide (CO) among WP smokers. Answers to these questions will help the FDA predict the impact of flavor regulation on WP experimentation and continued use. In this study, investigators will use clinical laboratory methods to answer these questions. Two groups of WP smokers will be recruited based on their use frequency: low (Beginners) vs. high frequency (Experienced) smokers (72/group; total 144; age 18-30). Each participant will undergo 2 WP smoking sessions that differ by flavor (preferred flavor; unflavored), while measurement of WP satisfaction, dependence, harm perception, and exposure to nicotine and toxicants will be conducted. The response of WP smokers at different stages of their WP smoking trajectory (Beginners vs. Experienced) to flavor manipulation, will allow to predict the effect of limiting flavors on a wide range of WP smokers. This project promises to provide the first evidence to guide the FDA in terms of the potential of regulating WP flavored tobacco on WP uptake and use in the US.

ELIGIBILITY:
Inclusion Criteria:

* Generally healthy individuals (determined by physical examination).
* Age of 18-30 years.
* Is willing to provide informed consent.
* Is willing to attend the lab as required by the study protocol.
* WP smokers who smoke flavored WP tobacco.
* Have abstained from WP for 12 hours prior to each session

Exclusion Criteria:

* Report smoking cigarettes regularly (> 5 cigarettes/month in the past year).
* Report regular use of any other tobacco/nicotine product (e.g., e-cig, pipes, cigars) in the past year.
* Women who are breast-feeding or test positive for pregnancy (by urinalysis at screening).
* Individuals with self-reported history of chronic disease or psychiatric conditions.
* Individuals with history of or active cardiovascular disease, low or high blood pressure, seizures, and regular use of prescription medications (other than vitamins or birth control).

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 144 (Actual)
Dates: Start 2017-03-21 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Plasma nicotine | During participants' 1st and 2nd visit. Blood will be taken 2 times in each smoking session: before and after an approximately 45-min ad lib use period
  Change in plasma nicotine level

SECONDARY OUTCOMES:
Puff topography | During participants' 1st and 2nd visit. Puffing behavior is continuously measured during each smoking session (an approximately 45-min ad lib use period)
  measurement of puffing behavior
Minnesota Nicotine Withdrawal Scale | During participants' 1st and 2nd visit. Questionnaire will be administered 2 times in each smoking session: before and after an approximately 45-min ad lib use period.
  This scale is used to assess the extent to which product use reduces tobacco abstinence symptoms, and consists of 11 items scored 0 - 100. These items are presented as Visual Analog Scale with item (measure) centered above a horizontal line anchored on the left with not at all and on the right with extremely.
Tiffany-Drobes Questionnaire of Smoking Urges | During participants' 1st and 2nd visit. Questionnaire will be administered 2 times in each smoking session: before and after an approximately 45-min ad lib use period.
  This scale is used to assess the extent to which product use reduces tobacco abstinence symptoms, and consists of 10 items that are scored 0 - 7. Rated on a 7-point Likert scale ranging from 0 (strongly disagree) to 6 (strongly agree).
Carbon monoxide levels | During participants' 1st and 2nd visit. Carbon monoxide levels will be measured 2 times in each smoking session:before and after an approximately 45-min ad lib use period
  Change in carbon monoxide levels (in parts per mission)
Harm perception | During participants' 1st and 2nd visit. Questionnaire will be administered after each of the 2 smoking sessions. Each session is approximately 45-min ad lib use period.
  This scale assess waterpipe harm perception and measure perceptions of waterpipe relative risk compared to cigarettes. The scale will be scored on a 7-point scale ranging from 1 (not at all harmful), to 7 (extremely harmful).
Duke Sensory Questionnaire | During participants' 1st and 2nd visit. Questionnaire will be administered after each of the 2 smoking sessions. Each session is approximately 45-min ad lib use period.
  This scale assess participants sensory experience of the inhaled product. The scale has nine items. All items will be scored on a 7-point Likert scale anchored at the extremes (1= not at all; 7=extremely).
The Cigarette/WP Evaluation Scale (WES) | During participants' 1st and 2nd visit. Questionnaire will be administered after each of the 2 smoking sessions. Each session is approximately 45-min ad lib use period.
  This scale assesses participants' perception of the smoked waterpipe, The scale has 11 items. All items will be scored on a 7-point Likert scale anchored at the extremes (1= not at all; 7=extremely).

OTHER OUTCOMES:
Heart rate | During participants' 1st and 2nd visit. Heat rate will be measured from baseline continuously throughout each approximately 45-min sessionr
  Change in heart rate, measured in beats per minute
Blood pressure | During participants' 1st and 2nd visit. Blood pressure will be measured from baseline continuously throughout each approximately 45-min session
  Change in blood pressure, measured in mm/hg

CONTACTS AND LOCATIONS:
Locations (1):
- Florida International University, Miami, Florida, United States